CLINICAL TRIAL: NCT03050762
Title: Comprehensive Data Collection and Follow-Up for Patients With Thyroid, Parathyroid and Adrenal Disease
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA11-0695
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Endocrine Disease
Keywords: Endocrine Disease; Thyroid disease; Parathyroid disease; Adrenal disease; Data Review; Database
MeSH Terms: conditions — Endocrine System Diseases; Thyroid Diseases; Parathyroid Diseases; Adrenal Gland Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endocrine Disease Group: Information from the medical record recorded and entered into a research database.
  Starting about 2-3 years after testing and/or diagnosis and/or treatment and continuing for up to 15 years after surgery, research team will contact participant by phone to follow up.
  Interventions: Other: Data Collection; Behavioral: Follow Up

INTERVENTIONS:
Other: Data Collection — Participant information collected from either source document or direct participant response.
Behavioral: Follow Up — Participants followed up at the return to clinic visits. If participant cannot come to clinic, either a questionnaire mailed requesting follow-up, or participant called. Participants followed for a length of 15 years at intervals of every 2-3 years.

SUMMARY:
The goal of this data review study is to collect data to learn more about thyroid, parathyroid, and adrenal disease.

DETAILED DESCRIPTION:
If participant or participant's child agrees to take part in this study, information from the medical record will be recorded and entered into a research database at MD Anderson. Researchers will use this data to learn more about participant's or participant's child's current or suspected illness, surgery, and/or recovery as well as participant's or participant's child's medical history.

Length of Study Participant's or participant's child's active participation on this study will be over after 15 years.

Follow-Up Phone Calls Starting about 2-3 years after participant's or participant's child's testing and/or diagnosis and/or treatment and continuing for up to 15 years after participant's surgery, a member of the research team will contact participant by phone to follow up and see how participant or participant's child are doing. The first time participant receives a phone call or are asked in the clinic, participant will be asked for participant's verbal consent for participant or, if this is for participant's child, on behalf of participant's child, to speak to the member of the research team before participant or participant's child are asked any questions. After participant agrees, participant or participant's child will be asked a series of questions related to participant's or participant's child's disease (takes about 20-30 minutes) that ask about participant's or participant's child's current medical status and medical history. Each phone call should take 20-30 minutes to complete.

If participant or participant's child are scheduled for a routine clinic visit around the time of participant's or participant's child's next follow-up phone call, the research team member may talk to participant or participant's child in person at that time, or a questionnaire can be mailed to participant or participant's child if needed.

This is an investigational study.

Up to 15,000 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients that are being seen at MD Anderson with diagnosed or suspected endocrine disease. Patients will be selected from patients undergoing evaluation and/or treatment in the Endocrine Center, either by selection from a participating Endocrine physician or by screening from study personnel for patients scheduled to be seen in the Endocrine Clinic.
2. In addition, we intend to contact family members of patients who are enrolled on the study, and found to be deceased at follow-up, to request permission to obtain cause of death, to determine whether cause of death may be related to endocrine disease.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants seen at MD Anderson Cancer Center with diagnosed or suspectied endocrine disease.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2011-10-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Research Database Compilation from Suspected or Diagnosed Endocrine Disease Participants by Medical Record Review and Follow Up | 15 years
  Database compiled from continuous collection of data on patients diagnosed with surgical endocrine disease or patients who are at risk for developing endocrine neoplasia and/or disease, and by prospective follow-ups of patient populations.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org